CLINICAL TRIAL: NCT00213135
Title: A Phase III, Randomized, Double-blind, Three-arm, Placebo-controlled, Multi-center Study to Evaluate the Safety and Efficacy of Oral Cladribine in Subjects With Relapsing-remitting Multiple Sclerosis (RRMS)
Brief Title: A Safety and Efficacy Study of Oral Cladribine in Subjects With Relapsing-remitting Multiple Sclerosis (RRMS)
Acronym: CLARITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25643
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Cladribine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- Cladribine 5.25 mg/kg (Experimental)
  Interventions: Drug: Cladribine 5.25 mg/kg
- Cladribine 3.5 mg/kg (Experimental)
  Interventions: Drug: Cladribine 3.5 mg/kg
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cladribine 5.25 mg/kg — Cladribine tablet will be administered as cumulative dose of 0.875 milligram per kilogram (mg/kg) over a course of 4 or 5 consecutive days of 28-day period at Week 1, 5, 9, 13, 48, and 52 resulting in total cladribine dose of 5.25 mg/kg during the treatment period of 96 weeks.
  Arms: Cladribine 5.25 mg/kg
Drug: Cladribine 3.5 mg/kg — Cladribine tablet will be administered as cumulative dose of 0.875 mg/kg over a course of 4 or 5 consecutive days of 28-day period at Weeks 1, 5, 48, and 52 and placebo matched to cladribine tablet will be administered at Week 9 and 13 resulting in total cladribine dose of 3.5 mg/kg during the treatment period of 96 weeks.
  Arms: Cladribine 3.5 mg/kg
Other: Placebo — Placebo matched to cladribine tablet will be administered over a course of 4 or 5 consecutive days of 28-day period at Weeks 1, 5, 9, 13, 48 and 52 during the treatment period of 96 weeks.
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if cladribine tablets are a safe and effective treatment for relapsing-remitting multiple sclerosis (RRMS).

DETAILED DESCRIPTION:
This is a randomized, double-blind, three-arm, placebo-controlled, multi-center study. The study includes a pre-study evaluation period (up to 28 days prior to the start of treatment); an initial treatment period from Week 1 to 48; and a re-treatment period during Week 49 to 96.

During the initial treatment period (Week 1 to 48), eligible subjects are equally randomized by a central randomization system to receive either a) cladribine at a low dose (0.875 milligram per kilogram per course [mg/kg/course] for two courses plus placebo for two courses); b) cladribine at a high dose (0.875 mg/kg/course for four courses); or c) placebo (four courses). During the re-treatment period (Weeks 49 to 96), subjects received either a) cladribine at a low dose (0.875 mg/kg/course for two courses); or b) placebo (two courses).

For all randomized subjects, there is a rescue option of treatment with Rebif® (interferon beta-1a 44 microgram (mcg) given subcutaneously three times a week), if the subject experienced more than one qualifying relapse, and/or experienced a sustained increase in their EDSS score of greater than or equal to (>=) 1 point, or >=1.5 points if baseline EDSS score is 0, (over a period of three months or greater), during a calendar year beginning at Week 24.

To maintain the blind, there is a treating physician who view clinical laboratory results and assess adverse events and safety information, and an independent blinded evaluating physician who will perform neurological exams. A central neuroradiology center, also blinded to treatment, will assess magnetic resonance imaging (MRI) evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 65 years of age (inclusive, at time of informed consent)
* Has definite MS according to the McDonald criteria
* Has relapsing-remitting disease with 1 or more relapses within 12 months prior to Study Day 1
* Must have been clinically stable and not has a relapse within 28 days prior to Study Day 1
* Has MRI consistent with MS at the pre-study evaluation according to the Fazekas criteria
* Has a EDSS score from 0 to 5.5, inclusive
* Weighed between 40-120 kilogram (kg), inclusive
* If female, she must:

  1. be post-menopausal or surgically sterilized; or
  2. uses a hormonal contraceptive, intra uterine device, diaphragm with spermicide, or condom with spermicide, for the duration of the study; and
  3. be neither pregnant nor breast-feeding
* If male, he must be willing to use contraception to avoid pregnancies
* Be willing and able to comply with study procedures for the duration of the study
* Voluntarily provides written informed consent, and for United states of America (USA) sites only, a subject authorization under Health Insurance Portability and Accountability Act (HIPAA)

Exclusion Criteria:

* Has secondary progressive MS (SPMS) or primary progressive MS (PPMS)
* Prior use of disease modifying drugs (DMDs) within the last 3 months, or 2 or more prior treatment failures with DMDs on the basis of efficacy
* Has significant leukopenia (white blood cell count less than 0.5 times the lower limit of normal of the central laboratory) within 28 days prior to Study Day 1
* Has received cladribine, mitoxantrone, total lymphoid irradiation, myelosuppressive therapy, campath-1h, cyclophosphamide, azathioprine, methotrexate or natalizumab
* Has received oral or systemic corticosteroids or adrenocorticotropic hormone within 28 days prior to Study Day 1
* Has compromised immune function or infection
* Has received oral or systemic corticosteroids or adrenocorticotropic hormone within 28 days prior to Study Day 1
* Has received cytokine-based therapy, intravenous immunoglobulin therapy, or plasmapheresis within 3 months prior to Study Day 1
* Has platelet and absolute neutrophil counts below the lower limit of normal range within 28 days prior to Study Day 1
* Has prior or current history of malignancy
* Has a history of persistent anemia, leukopenia, neutropenia, or thrombocytopenia after immunosuppressive therapy
* Has systemic disease that, in the opinion of the Investigator, might interfere with subject safety, compliance or evaluation of the condition under Study (for example, insulin-dependent diabetes, Lyme disease, clinically significant cardiac, hepatic, or renal disease, Human Immunodeficiency Virus, or Human T-Cell Lymphotrophic Virus Type-1)
* Has a psychiatric disorder that, in the opinion of the Investigator, was unstable or would preclude safe participation in the study
* Has allergy or hypersensitivity to gadolinium, to cladribine or any of its excipients
* Has used any investigational drug or experimental procedure within 6 months prior to Study Day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1326 (Actual)
Dates: Start 2005-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Greenberg, M.D., Study Director — EMD Serono

REFERENCES:
- [Result] Giovannoni G, Comi G, Cook S, Rammohan K, Rieckmann P, Soelberg Sorensen P, Vermersch P, Chang P, Hamlett A, Musch B, Greenberg SJ; CLARITY Study Group. A placebo-controlled trial of oral cladribine for relapsing multiple sclerosis. N Engl J Med. 2010 Feb 4;362(5):416-26. doi: 10.1056/NEJMoa0902533. Epub 2010 Jan 20. PMID 20089960
- [Derived] Stefano N, Sormani MP, Giovannoni G, Rammohan K, Leist TP, Coyle PK, Dangond F, Alexandri N, Galazka A. Relapses in people with multiple sclerosis treated with cladribine tablets followed for up to 5 years: a plain language summary. Neurodegener Dis Manag. 2022 Dec;12(6):303-310. doi: 10.2217/nmt-2022-0019. Epub 2022 Aug 26. PMID 36017797
- [Derived] Giovannoni G, Comi G, Rammohan K, Rieckmann P, Dangond F, Jack D, Vermersch P. Disease stability over five years in people with multiple sclerosis treated with cladribine tablets: a plain language summary. Neurodegener Dis Manag. 2022 Dec;12(6):295-301. doi: 10.2217/nmt-2022-0018. Epub 2022 Aug 26. PMID 36017780
- [Derived] Vermersch P, Galazka A, Dangond F, Damian D, Wong SL, Jack D, Harty G. The effect of cladribine tablets in people with more active multiple sclerosis: a plain language summary. Neurodegener Dis Manag. 2022 Dec;12(6):285-293. doi: 10.2217/nmt-2022-0009. Epub 2022 Aug 3. PMID 35920065
- [Derived] Oh J, Walker B, Giovannoni G, Jack D, Dangond F, Nolting A, Aldridge J, Lebson LA, Leist TP. Side effects that occurred early in people with multiple sclerosis during the first year of treatment with cladribine tablets: a plain language summary. Neurodegener Dis Manag. 2022 Feb 1;12(1):1-7. doi: 10.2217/nmt-2021-0041. Epub 2022 Jan 12. PMID 35019731
- [Derived] Giovannoni G, Coyle PK, Vermersch P, Walker B, Aldridge J, Nolting A, Galazka A, Lemieux C, Leist TP. Integrated Lymphopenia Analysis in Younger and Older Patients With Multiple Sclerosis Treated With Cladribine Tablets. Front Immunol. 2021 Dec 24;12:763433. doi: 10.3389/fimmu.2021.763433. eCollection 2021. PMID 35003076
- [Derived] Giovannoni G, Comi G, Rammohan K, Rieckmann P, Dangond F, Keller B, Jack D, Vermersch P. Long-Term Disease Stability Assessed by the Expanded Disability Status Scale in Patients Treated with Cladribine Tablets 3.5 mg/kg for Relapsing Multiple Sclerosis: An Exploratory Post Hoc Analysis of the CLARITY and CLARITY Extension Studies. Adv Ther. 2021 Sep;38(9):4975-4985. doi: 10.1007/s12325-021-01865-w. Epub 2021 Aug 9. PMID 34370275
- [Derived] De Stefano N, Sormani MP, Giovannoni G, Rammohan K, Leist T, Coyle PK, Dangond F, Keller B, Alexandri N, Galazka A. Analysis of frequency and severity of relapses in multiple sclerosis patients treated with cladribine tablets or placebo: The CLARITY and CLARITY Extension studies. Mult Scler. 2022 Jan;28(1):111-120. doi: 10.1177/13524585211010294. Epub 2021 May 10. PMID 33969750
- [Derived] Giovannoni G, Galazka A, Schick R, Leist T, Comi G, Montalban X, Damian D, Dangond F, Cook S. Pregnancy Outcomes During the Clinical Development Program of Cladribine in Multiple Sclerosis: An Integrated Analysis of Safety. Drug Saf. 2020 Jul;43(7):635-643. doi: 10.1007/s40264-020-00948-x. PMID 32447743
- [Derived] Terranova N, Hicking C, Dangond F, Munafo A. Effects of Postponing Treatment in the Second Year of Cladribine Administration: Clinical Trial Simulation Analysis of Absolute Lymphocyte Counts and Relapse Rate in Patients with Relapsing-Remitting Multiple Sclerosis. Clin Pharmacokinet. 2019 Mar;58(3):325-333. doi: 10.1007/s40262-018-0693-y. PMID 29992396
- [Derived] Afolabi D, Albor C, Zalewski L, Altmann DR, Baker D, Schmierer K. Positive impact of cladribine on quality of life in people with relapsing multiple sclerosis. Mult Scler. 2018 Oct;24(11):1461-1468. doi: 10.1177/1352458517726380. Epub 2017 Aug 17. PMID 28817997
- [Derived] Savic RM, Novakovic AM, Ekblom M, Munafo A, Karlsson MO. Population Pharmacokinetics of Cladribine in Patients with Multiple Sclerosis. Clin Pharmacokinet. 2017 Oct;56(10):1245-1253. doi: 10.1007/s40262-017-0516-6. PMID 28255849
- [Derived] De Stefano N, Giorgio A, Battaglini M, De Leucio A, Hicking C, Dangond F, Giovannoni G, Sormani MP. Reduced brain atrophy rates are associated with lower risk of disability progression in patients with relapsing multiple sclerosis treated with cladribine tablets. Mult Scler. 2018 Feb;24(2):222-226. doi: 10.1177/1352458517690269. Epub 2017 Jan 31. PMID 28140753
- [Derived] Ali S, Paracha N, Cook S, Giovannoni G, Comi G, Rammohan K, Rieckmann P, Sorensen PS, Vermersch P, Greenberg S, Scott DA, Joyeux A; CLARITY (CLAdRIbine Tablets treating multiple sclerosis orallY) Study Group. Reduction in healthcare and societal resource utilization associated with cladribine tablets in patients with relapsing-remitting multiple sclerosis: analysis of economic data from the CLARITY Study. Clin Drug Investig. 2012 Jan 1;32(1):15-27. doi: 10.2165/11593310-000000000-00000. PMID 22017519

RESULTS

PARTICIPANT FLOW:
Groups:
- Cladribine 5.25 mg/kg: Cladribine tablet administered as cumulative dose of 0.875 milligram per kilogram (mg/kg) over a course of 4 or 5 consecutive days of 28-day period at Week 1, 5, 9, 13, 48, and 52 resulting in total cladribine dose of 5.25 mg/kg during the treatment period of 96 weeks.
- Cladribine 3.5 mg/kg: Cladribine tablet administered as cumulative dose of 0.875 mg/kg over a course of 4 or 5 consecutive days of 28-day period at Week 1, 5, 48, and 52 and placebo matched to cladribine tablet was administered at Week 9 and 13 resulting in total cladribine dose of 3.5 mg/kg during the treatment period of 96 weeks.
- Placebo: Placebo matched to cladribine tablet administered over a course of 4 or 5 consecutive days of 28-day period at Week 1, 5, 9, 13, 48 and 52 during the treatment period of 96 weeks.
Period: Overall Study
Arm/Group | Cladribine 5.25 mg/kg | Cladribine 3.5 mg/kg | Placebo
Started | 456 | 433 | 437
Completed | 406 | 398 | 380
Not Completed | 50 | 35 | 57
Not completed — Adverse Event | 9 | 5 | 5
Not completed — Lost to Follow-up | 11 | 8 | 4
Not completed — Protocol Violation | 4 | 4 | 10
Not completed — Death | 1 | 1 | 2
Not completed — Disease progression | 4 | 5 | 21
Not completed — Other | 21 | 12 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cladribine 5.25 mg/kg | Cladribine 3.5 mg/kg | Placebo | Total
Number analyzed (Participants) | 456 | 433 | 437 | 1326
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.1 (9.9) | 37.9 (10.3) | 38.7 (9.9) | 38.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 312 | 298 | 288 | 898
  Male | 144 | 135 | 149 | 428

OUTCOME MEASURES:

1. Primary Outcome: Annualized Qualifying Relapse Rate
Description: A qualifying relapse was defined as an increase of 2 points in at least one functional system of the expanded disability status scale (EDSS) or an increase of 1 point in at least two functional systems (excluding changes in bowel or bladder function or cognition) in the absence of fever, lasting for at least 24 hours and to have been preceded by at least 30 days of clinical stability or improvement. Expanded disability status scale (EDSS) assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to multiple sclerosis [MS]) was calculated. The annualized relapse rate for each treatment group was calculated as the total number of confirmed relapses divided by the total number of days on study multiplied by 365.25.
Time Frame: Week 96
Population: The intention-to-treat (ITT) population included all participants who were randomized in the study.
Measure: Number (95% Confidence Interval); unit: relapses per year
Arm/Group | Cladribine 5.25 mg/kg | Cladribine 3.5 mg/kg | Placebo
Number analyzed (Participants) | 456 | 433 | 437
relapses per year | 0.15 (0.58) [0.12 to 0.17] | 0.14 (0.59) [0.12 to 0.17] | 0.33 (0.88) [0.29 to 0.38]
Statistical Analysis 1: Comparison: Cladribine 5.25 mg/kg vs Placebo; Test type: Superiority or Other; p < 0.001, Wald Chi-square test; Relative Risk = 0.43, 95% CI 2-sided [0.35 to 0.54], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Cladribine 3.5 mg/kg vs Placebo; Test type: Superiority or Other; p < 0.001, Wald Chi-square test; Relative Risk = 0.43, 95% CI 2-sided [0.34 to 0.54], Standard Error of Mean 0.12

2. Secondary Outcome: Percentage of Relapse-free Participants
Description: A qualifying relapse was defined as an increase of 2 points in at least one functional system of the EDSS or an increase of 1 point in at least two functional systems (excluding changes in bowel or bladder function or cognition) in the absence of fever, lasting for at least 24 hours and to have been preceded by at least 30 days of clinical stability or improvement. Expanded disability status scale (EDSS) assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated.
Time Frame: Week 96
Population: The ITT population included all participants who were randomized in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Cladribine 5.25 mg/kg | Cladribine 3.5 mg/kg | Placebo
Number analyzed (Participants) | 456 | 433 | 437
percentage of participants | 78.9 | 79.7 | 60.9

3. Secondary Outcome: Time to Disability Progression
Description: Time to disability progression was defined as the time to a sustained increase in EDSS score of at least 1 point if baseline EDSS score between 0.5 and 4.5 inclusively, or at least 1.5 points if the baseline EDSS score was 0, or at least 0.5 point if the baseline EDSS score was at least 5, over a period of at least three months. Expanded disability status scale (EDSS) assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. Tenth Percentile of time to sustained increase in EDSS score was reported using Kaplan-Meier survival curve.
Time Frame: Baseline up to Week 96
Population: The ITT population included all participants who were randomized in the study.
Measure: Number; unit: months
Arm/Group | Cladribine 5.25 mg/kg | Cladribine 3.5 mg/kg | Placebo
Number analyzed (Participants) | 456 | 433 | 437
months | 13.6 | 13.6 | 10.8

4. Secondary Outcome: Mean Number of Combined Unique (CU) Lesions, Active Time Constant 2 (T2) Lesions, and Active Time Constant 1 (T1) Gadolinium-Enhanced (Gd+) Lesions Per Participant Per Scan
Description: Mean Number of CU lesions, active T2 lesions, and active T1 Gd+ lesions were measured by using magnetic resonance imaging (MRI) scans.
Time Frame: Week 96
Population: The ITT population included all participants who were randomized in the study.
Measure: Least Squares Mean (Standard Error); unit: lesions
Arm/Group | Cladribine 5.25 mg/kg | Cladribine 3.5 mg/kg | Placebo
Number analyzed (Participants) | 456 | 433 | 437
lesions
  CU lesions | 0.38 (0.08) | 0.43 (0.08) | 1.72 (0.08)
  Active T1 Gd+ lesions | 0.11 (0.05) | 0.12 (0.05) | 0.91 (0.05)
  Active T2 lesions | 0.33 (0.06) | 0.38 (0.07) | 1.43 (0.06)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 96
Description: Safety population included all the randomized participants who received at least one dose of stud medication with follow-up safety data
Arm/Group | Cladribine 5.25 mg/kg | Cladribine 3.5 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 41/454 | 36/430 | 28/435
Other Adverse Events (participants affected / at risk) | 324/454 | 286/430 | 242/435
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine 5.25 mg/kg (N=454) | Cladribine 3.5 mg/kg (N=430) | Placebo (N=435)
Pneumonia (Infections and infestations) | 3 | 3 | 3
Adnexitis (Infections and infestations) | 2 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Actinomycosis (Infections and infestations) | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0
Endometritis (Infections and infestations) | 1 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Herpes zoster infection neurological (Infections and infestations) | 1 | 0 | 0
Herpes zoster oticus (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0
Myocarditis bacterial (Infections and infestations) | 0 | 0 | 1
Orchitis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis relapsing (Gastrointestinal disorders) | 0 | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 2 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 0 | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 0 | 1
Cardiac hypertrophy (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Drowning (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Facial spasm (Nervous system disorders) | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Nephrosclerosis (Renal and urinary disorders) | 0 | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0
Breast dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arterial disorder (Vascular disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cladribine 5.25 mg/kg (N=454) | Cladribine 3.5 mg/kg (N=430) | Placebo (N=435)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 27 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 34 | 28
Depression (Psychiatric disorders) | 25 | 18 | 13
Diarrhoea (Gastrointestinal disorders) | 31 | 30 | 29
Fatigue (General disorders) | 27 | 20 | 26
Headache (Nervous system disorders) | 94 | 104 | 75
Influenza (Infections and infestations) | 34 | 27 | 27
Influenza like illness (General disorders) | 27 | 34 | 31
Insomnia (Psychiatric disorders) | 14 | 25 | 17
Leukopenia (Blood and lymphatic system disorders) | 39 | 23 | 3
Lymphocyte count decreased (Investigations) | 26 | 13 | 0
Lymphopenia (Blood and lymphatic system disorders) | 142 | 92 | 8
Nasopharyngitis (Infections and infestations) | 58 | 62 | 56
Nausea (Gastrointestinal disorders) | 49 | 43 | 39
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 16 | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 | 19 | 25
Upper respiratory tract infection (Infections and infestations) | 52 | 54 | 42
Urinary tract infection (Infections and infestations) | 32 | 23 | 39
Vertigo (Ear and labyrinth disorders) | 23 | 14 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other